CLINICAL TRIAL: NCT03756896
Title: Maintenance Therapy With Carfilzomib, Pomalidomide and Dexamethasone (CPd) in High-Risk Myeloma Patients: A Phase 2 Study With a Safety Run-In
Brief Title: Carfilzomib, Pomalidomide, and Dexamethasone in Treating Patients With High-Risk Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Amgen (Industry); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ajay Nooka, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00097882; NCI-2017-02052 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4101-17 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Dexamethasone; Calcium Dobesilate; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carfilzomib, pomalidomide, dexamethasone (Experimental): Patients receive carfilzomib IV over 30 minutes on days 1, 8, and 15, pomalidomide PO daily on days 1-21, and dexamethasone PO daily on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Drug: Pomalidomide

INTERVENTIONS:
Drug: Carfilzomib — Given IV
  Other Names: Kyprolis; PR-171
Drug: Dexamethasone — Given PO
  Other Names: Decadron; Dekacort; Dexameth; Hexadrol
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC-4047; Imnovid; Pomalyst

SUMMARY:
This phase II trial studies how well carfilzomib, pomalidomide, and dexamethasone work in treating patients with high-risk multiple myeloma. Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as pomalidomide and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving carfilzomib, pomalidomide, and dexamethasone may work better in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the ≥ complete response (CR) rates with carfilzomib, pomalidomide and dexamethasone (CPd) maintenance.

SECONDARY OBJECTIVES:

I. To determine the improved progression free survival (PFS) with CPd maintenance among high-risk patients.

II. To determine the best response rates (very good partial response rate [VGPR], stringent complete response [sCR] rate) with CPd maintenance.

II. To evaluate the safety of the CPd combination as maintenance regimen.

III. To characterize safety in subjects who receive CPd maintenance.

IV. To evaluate the duration of response (DOR).

V. To evaluate the overall survival (OS) in high-risk patients.

VI. To evaluate the minimal residual disease (MRD) detection with CPd maintenance.

OUTLINE:

Patients receive carfilzomib intravenously (IV) over 30 minutes on days 1, 8, and 15, pomalidomide orally (PO) daily on days 1-21, and dexamethasone PO daily on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the following criteria on screening examination to be eligible to participate in the study; all laboratory assessments should be performed within 28 days of initiation of protocol therapy unless otherwise specified; subject is, in the investigator's opinion, willing and able to comply with the protocol requirements
* Subject has given voluntary signed written informed consent before performance of any study-related procedure that is not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to their future medical care
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1
* Subject is a transplant-eligible patient that have undergone autologous stem cell transplant (ASCT) within one year of their diagnosis and have achieved ≥ partial response (PR) based on International Myeloma Working Group (IMWG) standard criteria
* Patients with high risk disease defined as

  * Presence of del(17p); t(4;14); t(14;16); t(14;20) by fluorescence in situ hybridization (FISH) or by cytogenetics (CTG)
  * Plasma cell leukemia at diagnosis with ≥ 20% circulating plasma cells on peripheral blood
* Subject agrees to refrain from blood donations during therapy on study and for 90 days after therapy is completed
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 milli-International units (mIU)/mL within 10-14 days prior to and again within 24 hours of starting pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking pomalidomide through 90 days after the last dose of study drug; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy from the time of signing the informed consent form through 90 days after the last dose of study drug; all patients must be registered in and must comply with all requirements of the pomalidomide Risk Evaluation and Mitigation Strategies (REMS) program; male subjects should refrain from sperm donation for at least 90 days after the last dose of carfilzomib or pomalidomide

  * FCBP refers to sexually mature female, regardless of sexual orientation or whether they have undergone tubal ligation, who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally menopausal for at least 24 consecutive months

Exclusion Criteria:

* Diagnosed with smoldering multiple myeloma (MM), monoclonal gammopathy of undetermined significance, Waldenstrom's macroglobulinemia, polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome, amyloidosis or standard risk myeloma or secondary plasma cell leukemia
* High risk patients that did not achieve ≥ PR after stem cell transplant
* Participant has ≥ grade 2 peripheral neuropathy on clinical examination within 21 days before initiation of protocol therapy
* Creatinine clearance < 30 mL/min (either actual or calculated value), within 21 days of initiation of protocol therapy; the Cockcroft-Gault formula should be used for calculating creatinine clearance values
* Platelet count < 75,000 cells/mm³ at time of screening evaluation; transfusion may not be used to meet platelet eligibility criteria within 7 days of obtaining screening evaluation
* Participants with an absolute neutrophil count (ANC) < 1000 cells/mm³ at time of screening evaluation; growth factors may not be used to meet ANC eligibility criteria within 14 days of obtaining screening evaluation
* Participants with hemoglobin level < 8.0 g/dL, at time of screening; transfusion may not be used to meet eligibility criteria within 7 days of obtaining screening evaluation
* Bilirubin > 1.5 x institutional upper limit of normal (ULN), within 21 days of initiation of protocol therapy
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]), alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]), or alkaline phosphatase > 3 x institutional ULN, within 21 days of initiation of protocol therapy
* Other ongoing or prior anti-myeloma therapy; patients may be receiving concomitant therapy with bisphosphonates and low dose corticosteroids (e.g., prednisone up to but no more than 10 mg p.o. once daily [q.d.] or its equivalent) for symptom management and comorbid conditions; doses of corticosteroid should be stable for at least 7 days prior to study treatment)
* Known significant cardiac abnormalities including:

  * Congestive heart failure, New York Heart Association (NYHA) class III or IV
  * Uncontrolled angina, arrhythmia or hypertension
  * Myocardial infarction within the past six months
  * Any other uncontrolled or severe cardiovascular condition
  * Prior cerebrovascular event with residual neurologic deficit
* Serious, intercurrent illness including, but not limited to, clinically relevant active infection, known active hepatitis B or C viral infection, known human immunodeficiency virus (HIV) infection, uncontrolled diabetes mellitus, or serious co-morbid medical conditions such as chronic restrictive pulmonary disease, and cirrhosis
* Any condition, including laboratory abnormalities, that in the opinion of the investigator places the subject at unacceptable risk if he/she were to participate in the study
* Prior malignancy (within the last 5 years) except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
* Known hypersensitivity to acyclovir or similar anti-viral drug
* Known intolerance to steroid therapy
* Contraindication or prior intolerance to thromboembolic prophylaxis with aspirin, warfarin or low-molecular weight heparin
* Participants with known central nervous system (CNS) disease
* Poor tolerability or known allergy to any of the study drugs or compounds of similar chemical or biologic composition to dexamethasone, boron or mannitol
* Female participants pregnant or breast-feeding
* Participants who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of the surgery
* Participants with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2025-06-24 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
≥ Complete response (CR) rates | Up to 2 years after study start
  Completed response (CR) rates will be determined for CPd maintenance.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From first dose until documented progression or death, assessed at 18 months
  Progression-free survival (PFS) is defined as the time from first dose until documented progression or death. A subject who neither progresses nor dies will be censored on the date of his or her last tumor assessments. PFS will be determined by using all enrolled patients in accordance with the intention to treat (ITT) principle.
Best response on-study | Up to 2 years after study start
  Best response on-study refers to the best response (very good partial response rate [VGPR], stringent complete response [sCR] rate) prior to discontinuation of all study therapy.
Objective response rate (ORR) defined as the proportion of treated subjects who achieve a best response of CR, stringent complete response (sCR), very good partial response (VGPR), or partial response (PR) | Up to 2 years after study start
  The objective response rate (ORR) will be assessed using International Myeloma Working Group (IMWG) criteria.
Duration of response (DOR) | From first response (PR or better) until a progression event (documented progression or death), assessed up to 2 years
  Duration of response (DOR) is the time from first response (PR or better) until a progression event (documented progression or death). Only subjects who ever achieved a response of PR or better will be considered. Subjects who neither progress nor die will be censored on the date of their last tumor assessment.
Overall survival (OS) | Up to 2 years after study start
  Overall survival (OS) is defined as the time from first dose until documented death.
Minimal residual disease (MRD) detection | Up to 2 years after study start
  The achievement of minimal residual disease (MRD) will be evaluated and reported on patients that achieve a complete response. MRD testing will be performed by adaptive clonoSEQ testing.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Nooka, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT03756896/ICF_000.pdf